CLINICAL TRIAL: NCT05535764
Title: Allogeneic Hematopoietic Cell Transplantation With Pegylated Interferon Alfa-2a for Primary and Secondary Myelofibrosis (ATIOM)
Brief Title: Allogeneic Hematopoietic Cell Transplantation With Pegylated Interferon Alfa-2a for Primary and Secondary Myelofibrosis
Acronym: ATIOM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI149616
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): A 3+3 dose de-escalation design will be used to determine the recommended phase 2 dose,while ensuring the safety and tolerability of the treatment. In this trial, the dose determined to be the maximum tolerated dose will be the recommended phase 2 dose and will be utilized in the cohort expansion.
  Interventions: Drug: Pegylated interferon alpha2a

INTERVENTIONS:
Drug: Pegylated interferon alpha2a — PegINFa will be given once every 2 weeks by subcutaneous administration in the abdomen or thigh.

SUMMARY:
This is a single site, open-label, dose de-escalation, Phase 1 study of pegylated interferon alfa-2a administered after alloHCT in subjects with primary or secondary myelofibrosis. Part 1 of the study will assess the rate of dose-limiting toxicities (DLTs) during the DLT evaluation period and identify the Recommended Phase 2 Dose (RP2D). Once the RP2D is identified, 6 additional patients will be enrolled in the expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

Pre-Transplant Inclusion Criteria (Step 1)

* Male or female subject aged ≥ 18 years.
* Diagnosis of primary or secondary myelofibrosis.
* Eligible to undergo a myeloablative or reduced intensity conditioning regimen (MAC or RIC)
* Eligible to undergo a standard of care bone marrow biopsy with aspirate as part of his or her routine pre-transplant work-up.
* Peripheral blood stem cell (PBSC) graft
* 10/10 HLA matched related or matched unrelated donor
* ECOG performance status ≤ 2.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1.

Treatment Inclusion Criteria (Step 2)

* Male or female subject aged ≥ 18 years.
* Diagnosis of primary or secondary myelofibrosis.
* Have undergone a myeloablative or reduced-intensity conditioning regimen (MAC or RIC) and be 50-80 days from Day 0 of transplant at initiation of study therapy.
* Peripheral blood stem cell (PBSC) graft
* 10/10 HLA matched related or matched unrelated donor
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
    * TSH and T4 within normal limits or adequately controlled thyroid function.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1.
* Male subjects must agree to use a condom during intercourse for the duration of study therapy as described in Section 5.4.1.
* Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

Exclusion Criteria (Step 2)

* Receiving other investigational agents concurrently
* Prior systemic anti-cancer therapy or any investigational therapy within five half-lives prior to starting study treatment.
* Prior radiotherapy within 6 weeks prior to the first dose of study treatment.
* Major surgery within 6 weeks prior to starting study drug or patients who have not fully recovered from major surgery.
* The diagnosis of another malignancy within ≤ 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, or low-grade prostate cancer with Gleason Score ≤ 6).
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Graft-versus-host disease:

    ---Acute or chronic
  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
    * QTc prolongation defined as a QTcF > 500 ms.
    * Known congenital long QT.
    * Left ventricular ejection fraction < 55%.
    * Uncontrolled hypertension defined as ≥ 140/90 as assessed from the mean of three consecutive blood pressure measurements taken over 10 minutes.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Active infection including HIV, tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice) or hepatitis C.
* Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
* Autoimmune hepatitis or decompensated hepatic disease
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.5.1. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.
* History of neuropsychiatric disease, autoimmune disease, or pancreatitis.
* Presence of active interstitial lung disease or pneumonitis, bronchiolitis obliterans, pulmonary hypertension, ulcerative and hemorrhagic/ischemic colitis, and ophthalmologic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) during the DLT evaluation period | Start of treatment to 86 days after treatment initiation
  To identify the Recommended Phase 2 Dose (RP2D) of pegylated interferon alfa-2a in subjects undergoing allogeneic hematopoietic cell transplantation for primary or secondary myelofibrosis

SECONDARY OUTCOMES:
Assess the safety of pegylated interferon alfa-2a in the study population. | 3 years
  Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE version 5.0), seriousness, duration, and relationship to study treatment.
Assess the tolerability of pegylated interferon alfa-2a in the study population. | 3 years
  Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE version 5.0), seriousness, duration, and relationship to study treatment.
Assess the rate of treatment-related mortality in the study population. | 3 years
  Rate of treatment-related mortality which is defined as proportion of deaths in patients who have received at least one dose of study therapy, which is attributed to complications from alloHCT or conditioning therapy (in the absence of myelofibrosis relapse) from 30 days after the end of conditioning therapy to one week after the last dose of study therapy.
Assess leukemia-free survival (LFS) in the study population. | 3 years
  Rate of Leukemia-free survival (LFS) as defined from the day of allogeneic hematopoietic cell transplantation to the time documented disease relapse/progression (date of bone marrow blast count of 20% or greater or date of first peripheral blast count of 20% or greater that was subsequently confirmed to sustain for at least 8 weeks), initiation of non-protocol MF therapy, loss to follow-up, study end, or death from any cause, whichever comes first.
Assess the incidence of acute and/or chronic graft versus host disease (GVHD) in the study population | 3 years
  Cumulative incidence of Glucksberg grade II, III, and IV acute GVHD and incidence of mild, moderate or severe chronic GVHD per NIH grading criteria.
Assess Objective Response Rate (ORR) in the study population. | 3 Years
  Response rates according to IWG-MRT including, CR, PR, CI, PD, SD, or Relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Patel, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No